CLINICAL TRIAL: NCT03999554
Title: Phase 1b Clinical Study to Investigate the Safety and Immunogenicity of the Bris10 (A/Brisbane/10/2007) M2SR and Sing2016 (A/Singapore/INFIMH-16-0019/2016) M2SR H3N2 Monovalent Influenza Vaccines
Brief Title: Safety and Immunogenicity of the Bris10 M2SR and Sing2016 M2SR H3N2 Monovalent Influenza Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FluGen Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: FLUGEN-H3N2-V003
Record Dates: First submitted 2019-06-18; First posted 2019-06-26 (Actual); Results first posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Influenza A

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled Phase 1 study evaluating the safety and immunogenicity of the Bris10 M2SR and Sing2016 M2SR H3N2 influenza vaccines delivered intranasally to healthy adults. Eligible subjects will be screened and randomized to receive two administrations 28 days apart of Sing2016 M2SR at three dose levels, Bris10 M2SR at one dose level, or placebo in a 1:1:1:1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Low dose Sing2016 M2SR (Experimental): Low dose Sing2016 M2SR will be administered intranasally on days 1 and 29
  Interventions: Biological: LD Sing2016 M2SR H3N2 influenza vaccine
- Medium dose Sing2016 M2SR (Experimental): Medium dose Sing2016 M2SR will be administered intranasally on days 1 and 29
  Interventions: Biological: MD Sing2016 M2SR H3N2 influenza vaccine
- High dose Sing2016 M2SR (Experimental): High dose Sing2016 M2SR will be administered intranasally on days 1 and 29
  Interventions: Biological: HD Sing2016 M2SR H3N2 influenza vaccine
- Low dose Bris10 M2SR (Active Comparator): Low dose Bris10 M2SR will be administered intranasally on days 1 and 29
  Interventions: Biological: LD Bris10 M2SR H3N2 influenza vaccine
- Placebo (Placebo Comparator): Saline will be administered intranasally on days 1 and 29
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: LD Sing2016 M2SR H3N2 influenza vaccine — This group will receive a low dose of the Sing2016 M2SR H3N2 monovalent influenza vaccine administered intranasally.
  Arms: Low dose Sing2016 M2SR
Biological: MD Sing2016 M2SR H3N2 influenza vaccine — This group will receive a medium dose of the Sing2016 M2SR H3N2 monovalent influenza vaccine administered intranasally.
  Arms: Medium dose Sing2016 M2SR
Biological: HD Sing2016 M2SR H3N2 influenza vaccine — This group will receive a high dose of the Sing2016 M2SR H3N2 monovalent influenza vaccine administered intranasally.
  Arms: High dose Sing2016 M2SR
Biological: LD Bris10 M2SR H3N2 influenza vaccine — This group will receive a low dose of the Bris10 M2SR H3N2 monovalent influenza vaccine administered intranasally.
  Arms: Low dose Bris10 M2SR
Other: Placebo — This group will receive saline placebo administered intranasally.
  Arms: Placebo

SUMMARY:
This is a Phase I double-blind, randomized, placebo-controlled study in 250 healthy adults, 18-49 years of age, inclusive, who are in good health and meet all eligibility criteria. The purpose of this dose escalation clinical study is to assess the safety, tolerability/reactogenicity, and immunogenicity of H3N2 M2SR investigational vaccines for prevention of influenza, when delivered at higher dosages or in two doses . Eligible subjects will be screened and randomized to receive two administrations 28 days apart of Sing2016 M2SR at three dose levels (low, medium, high), Bris10 M2SR at one dose level (low), or placebo in a 1:1:1:1:1 ratio. Study duration will be approximately 8 months with subject participation duration approximately 7 months. The primary study objective is to assess the safety and reactogenicity of a monovalent live single replication influenza H3N2 M2SR vaccine.

DETAILED DESCRIPTION:
This is a Phase I double-blind, randomized, placebo-controlled study in 250 healthy adults, 18-49 years of age, inclusive, who are in good health and meet all eligibility criteria. This dose escalation clinical study is designed to assess the safety, tolerability/reactogenicity, and immunogenicity of H3N2 M2SR investigational vaccines for prevention of influenza, when delivered at increasing dosages or in two doses. Subjects will be enrolled in five groups in a 1:1:1:1:1 ratio. Arm 1 will receive a low dose of Sing2016 M2SR intranasally on days 1 and 29. Arm 2 will receive a medium dose of Sing2016 M2SR intranasally on days 1 and 29. Arm 3 will receive a high dose of Sing2016 M2SR intranasally on days 1 and 29. Arm 4 will receive a low dose of Bris16 M2SR intranasally on days 1 and 29. Arm 5 will receive a placebo intranasally on days 1 and 29. Study duration will be approximately 8 months with subject participation duration approximately 7 months. The primary study objective is to assess the safety and reactogenicity of a monovalent live single replication influenza H3N2 M2SR vaccine. The secondary study objectives are to evaluate systemic and mucosal immune responses induced by H3N2 M2SR vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Give written informed consent to participate.
2. Age 18 - 49 years old.
3. Judged suitable by the PI, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations.
4. Willing to use oral, implantable, transdermal or injectable contraceptives, or sexual abstinence, from screening and until 28 days after second vaccine dose.
5. Willing to adhere to the requirements of the study and willing and able to communicate with the Investigator and understand the requirements of the study.

Exclusion Criteria:

1. Abnormal screening hematology or chemistry value per the FDA Toxicity Guidance.
2. Pulse rate or blood pressure outside the reference range for this study population and considered as clinically significant by the Investigator.
3. Has an acute or chronic medical condition or history of a medical condition that, in the opinion of the Investigator, would render the study procedures unsafe or would interfere with the evaluation of the responses.
4. Presence or clinically significant history of lung disease, asthma, chronic obstructive pulmonary disease (COPD), or otherwise poor lung function.
5. Any confirmed or suspected immunosuppressive or immunodeficient state.
6. Presence of household member or close personal or professional (i.e., healthcare worker) who is a child under one year of age; is pregnant; has known immunodeficiency or is receiving immunosuppressant medication; is undergoing or soon to undergo cancer chemotherapy; has been diagnosed with emphysema, COPD, or other severe lung disease and resides in a nursing home; and/or has received a bone marrow or solid organ transplant.
7. Females who are pregnant or lactating.
8. Acute febrile illness within 72 hours prior to vaccination.
9. Any condition, in the opinion of the Investigator, (such as subjects who have medically high-risk conditions) that might interfere with the primary study objectives for safety of the study subject.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamuk Bilsel, Study Director — FluGen Inc; Carlos Fierro, MD, Principal Investigator — JCCT
Locations (4):
- United States (4):
  - RCA, Hollywood, Florida
  - JCCT, Lenexa, Kansas
  - AMR Lexington, Lexington, Kentucky
  - AMR Norfolk, Norfolk, Virginia

REFERENCES:
- [Derived] Eiden J, Fierro C, Schwartz H, Adams M, Ellis KJ, Aitchison R, Herber R, Hatta Y, Marshall D, Moser MJ, Belshe R, Greenberg H, Coelingh K, Kawaoka Y, Neumann G, Bilsel P. Intranasal M2SR (M2-Deficient Single Replication) H3N2 Influenza Vaccine Provides Enhanced Mucosal and Serum Antibodies in Adults. J Infect Dis. 2022 Dec 28;227(1):103-112. doi: 10.1093/infdis/jiac433. PMID 36350017

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Low Dose Bris10 M2SR | Placebo
Started | 42 | 41 | 40 | 42 | 41
Completed | 36 | 34 | 28 | 35 | 32
Not Completed | 6 | 7 | 12 | 7 | 9
Not completed — Lost to Follow-up | 4 | 5 | 4 | 5 | 8
Not completed — Protocol Violation | 0 | 0 | 5 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 2 | 1 | 1
Not completed — failure to comply with protocol requirements | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Low Dose Bris10 M2SR | Placebo | Total
Number analyzed (Participants) | 42 | 41 | 40 | 42 | 41 | 206
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 41 | 40 | 42 | 41 | 206
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 29 | 35 | 31 | 146
  Male | 17 | 15 | 11 | 7 | 10 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 16 | 18 | 20 | 18 | 96
  Not Hispanic or Latino | 18 | 25 | 22 | 22 | 23 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 7 | 6 | 7 | 11 | 35
  White | 36 | 34 | 34 | 33 | 29 | 166
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local and Systemic Adverse Events (AEs) Through 29 Days Post-vaccination With Bris10 M2SR and Cumulatively Through Day 209
Description: Record adverse events following one and two administrations of the Bris10 M2SR influenza vaccine to determine the number and percentage of study participants who experience any vaccine associated adverse events (AEs) or serious adverse events (SAEs) after Bris10 M2SR or placebo administration.
Time Frame: From baseline through study completion (Day 209)
Population: Study participants who received at least one inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Bris10 M2SR | Placebo
Number analyzed (Participants) | 42 | 41
Participants | 28 | 24

2. Primary Outcome: Number of Participants With Local and Systemic Adverse Events (AEs) Through 29 Days Post-vaccination With Sing2016 M2SR and Cumulatively Through Day 209
Description: Record adverse events following one and two administrations of the Sing2016 M2SR influenza vaccine to determine the number and percentage of study participants who experience any vaccine associated adverse events (AEs) or serious adverse events (SAEs) after Sing2016 M2SR or placebo administration.
Time Frame: From baseline through study completion (Day 209)
Population: Study participants who received at least one inoculation were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Placebo
Number analyzed (Participants) | 42 | 41 | 40 | 41
Participants | 26 | 29 | 30 | 24

3. Secondary Outcome: Percentage of Bris10 M2SR Subjects Demonstrating Seroconversion to Vaccine HA
Description: Assess the humoral immunogenicity of one administration of Bris10 M2SR vaccine to Bris 10 by HAI at day 29.
Time Frame: From baseline through 28 days post-dose 1 (Day 29)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Bris10 M2SR | Placebo
Number analyzed (Participants) | 38 | 38
Percentage of subjects | 28.9 [15.4 to 45.9] | 10.5 [2.9 to 24.8]

4. Secondary Outcome: Percentage of Sing2016 M2SR Subjects Demonstrating Seroconversion to Vaccine HA
Description: Assess the humoral immunogenicity of one administration of Sing2016 M2SR vaccine to Sing2016 by HAI at day 29
Time Frame: From baseline through 28 days post-dose 1 (Day 29)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Placebo
Number analyzed (Participants) | 40 | 38 | 31 | 38
Percentage of participants | 27.5 [14.6 to 43.9] | 36.8 [21.8 to 54] | 71.0 [52 to 85.8] | 0 [0 to 9.3]

5. Secondary Outcome: Percentage of Bris10 M2SR Subjects Demonstrating Seroconversion to Vaccine HA
Description: Assess the humoral immunogenicity of two administrations of Bris10 M2SR vaccine to Bris 10 by HAI at d57.
Time Frame: From baseline through 28 days post-dose 2 (Day 57)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Bris10 M2SR | Placebo
Number analyzed (Participants) | 37 | 35
Percentage of subjects | 40.5 [24.8 to 57.9] | 14.3 [4.8 to 30.3]

6. Secondary Outcome: Percentage of Sing2016 M2SR Subjects Demonstrating Seroconversion to Vaccine HA
Description: Assess the humoral immunogenicity of two administrations of Sing2016 M2SR vaccine to Sing2016 by HAI at day 57
Time Frame: From baseline through 28 days post-dose 2 (Day 57)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Placebo
Number analyzed (Participants) | 38 | 36 | 31 | 35
Percentage of subjects | 47.4 [31 to 64.2] | 55.6 [38.1 to 72.1] | 80.6 [62.5 to 92.5] | 0 [0 to 10]

7. Secondary Outcome: Percentage of Bris10 M2SR Subjects Demonstrating Mucosal Responses to Vaccine HA
Description: Assess the mucosal immunogenicity of one administration of Bris10 M2SR vaccine to Bris 10 by ELISA at day 29.
Time Frame: From baseline through 28 days post-dose 1 (Day 29)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Bris10 M2SR | Placebo
Number analyzed (Participants) | 36 | 36
Percentage of subjects | 22.2 [10.1 to 39.2] | 25.0 [12.1 to 42.2]

8. Secondary Outcome: Percentage of Bris10 M2SR Subjects Demonstrating Mucosal Responses to Vaccine HA
Description: Assess the mucosal immunogenicity of two administrations of Bris10 M2SR vaccine to Bris 10 by ELISA at day 57.
Time Frame: From baseline through 28 days post-dose 2 (Day 57)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Bris10 M2SR | Placebo
Number analyzed (Participants) | 33 | 31
Percentage of subjects | 39.4 [22.9 to 57.9] | 25.8 [11.9 to 44.6]

9. Secondary Outcome: Percentage of Sing2016 M2SR Subjects Demonstrating Mucosal Responses to Vaccine HA
Description: Assess the mucosal immunogenicity of two administrations of Sing2016 M2SR vaccine to Sing2016 by ELISA at day 57
Time Frame: From baseline through 28 days post-dose 2 (Day 57)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Placebo
Number analyzed (Participants) | 35 | 33 | 28 | 31
Percentage of subjects | 20 [8.4 to 36.9] | 45.5 [28.1 to 63.6] | 60.7 [40.6 to 78.5] | 19.4 [7.5 to 37.5]

10. Secondary Outcome: Percentage of Sing2016 M2SR Subjects Demonstrating Mucosal Responses to Vaccine HA
Description: Assess the mucosal immunogenicity of one administration of Sing2016 M2SR vaccine to Sing2016 by ELISA at day 29
Time Frame: From baseline through 28 days post-dose 1 (Day 29)
Population: Study subjects who received at least one inoculation were included.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Placebo
Number analyzed (Participants) | 38 | 36 | 29 | 36
Percentage of subjects | 15.8 [6.0 to 31.3] | 22.2 [10.1 to 39.2] | 37.9 [20.7 to 57.7] | 19.4 [8.2 to 36.0]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously from first administration of IP until study day 57. SAEs were collected until study day 209.
Description: Administration site and solicited AEs were recorded through 7 days after each vaccination (Days 8 and 29), unsolicited AEs were recorded through 28 days after the last vaccination (Day 57) and SAEs were recorded until Day 209.
Arm/Group | Low Dose Sing2016 M2SR | Medium Dose Sing2016 M2SR | High Dose Sing2016 M2SR | Low Dose Bris10 M2SR | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41 | 0/40 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41 | 0/40 | 0/42 | 1/41
Other Adverse Events (participants affected / at risk) | 26/42 | 29/41 | 30/40 | 28/42 | 24/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Sing2016 M2SR (N=42) | Medium Dose Sing2016 M2SR (N=41) | High Dose Sing2016 M2SR (N=40) | Low Dose Bris10 M2SR (N=42) | Placebo (N=41)
papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — metastatic papillary thyroid carcinoma, study day 125, not considered treatment emergent
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Sing2016 M2SR (N=42) | Medium Dose Sing2016 M2SR (N=41) | High Dose Sing2016 M2SR (N=40) | Low Dose Bris10 M2SR (N=42) | Placebo (N=41)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 9 | 15 | 13 | 14
cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 10 | 5 | 6
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 12 | 8 | 10
throat irritation (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 5 | 4 | 6
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 8 | 7 | 3
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 3 | 2
upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1
nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 1 | 1
nasal pruritis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 0
fatigue (General disorders) | 13 | 8 | 10 | 14 | 8
pyrexia (General disorders) | 5 | 3 | 3 | 1 | 1
headache (Nervous system disorders) | 12 | 9 | 11 | 14 | 10
myalgia (Musculoskeletal and connective tissue disorders) | 9 | 6 | 9 | 7 | 4
arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 3 | 2 | 3
nausea (Gastrointestinal disorders) | 4 | 1 | 2 | 2 | 5
AAT increase (Investigations) | 2 | 0 | 0 | 0 | 0
blood creatinine phosphate increase (Investigations) | 1 | 2 | 0 | 1 | 1
blood urine (Investigations) | 0 | 0 | 2 | 0 | 0
white blood cell increase (Investigations) | 0 | 2 | 0 | 0 | 0
bradycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 0
hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR has exclusive right to publish and authorize study publications or communications. INVESTIGATOR makes no presentations/publications of the Study or its results without prior SPONSOR review and approval. SPONSOR will have 90 days to request amendments including but not limited to details that may be detrimental to its intellectual property interests or to the conduct, completion, or analysis of the results of the Study by SPONSOR or its affiliates.

DOCUMENTS (2):
  • Study Protocol (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03999554/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/54/NCT03999554/SAP_001.pdf